CLINICAL TRIAL: NCT05437653
Title: Developing Magnetic Resonance Imaging Techniques to Explore the Brain-gut Axis to Food Intake in People With Obesity and Healthy Weight Participants
Brief Title: MRI Based Study to Assess Brain-gut Axis in Obesity
Acronym: BGImaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19047
Record Dates: First submitted 2022-04-08; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Obesity
Keywords: obesity; brain-gut axis; functional magnetic resonance imaging; gastric emptying; small bowel water content; high fat meal; carbohydrate meal; Blood-oxygen-level-dependent; cerebral blood flow; resting state fMRI
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Randomised parallel trial in human volunteers. Control (normal weight) group VS Obese group and High fat drink VS iso-caloric, iso-viscous Carbohydrate drink
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blinded study, and the study participant and assessor will be unaware of the nature of the drink. Subjects will be invited into 2 MRI scan visits to investigate the brain and gut responses (brain-gut axis) to a high fat drink and a carbohydrate drink. Drinks will be randomised across participants using research randomizer software (https://www.randomizer.org/).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Healthy weight group ( same age and sex)
  Interventions: Other: Nutritional Drink A; Other: Nutritional Drink B
- Obese group (Active Comparator): Obese group
  Interventions: Other: Nutritional Drink A; Other: Nutritional Drink B

INTERVENTIONS:
Other: Nutritional Drink A — 300 mL of a 22% high fat emulsion (Rapeseed oil, water, emulsifier)
Other: Nutritional Drink B — 300 mL of isocaloric, iso-volumetric and iso-viscous carbohydrate drink (maltodextrin)

SUMMARY:
The mechanism of neural communication between the brain and gut in the regulation of food intake is complex and not fully understood. Magnetic Resonance Imaging (MRI) is a powerful non-invasive imaging tool that allows studying the function of the brain and gut. The aim of this study is to develop MRI methods to combine brain and gut imaging in a single MRI scan session. The developed techniques will then be used to assess the brain-gut axis to a high fat drink compared with iso-caloric/iso-viscous/iso-volumetric carbohydrate drink in people with obesity and healthy weight participants. The findings could provide a possible explanation for why some people are heavier than others.

DETAILED DESCRIPTION:
20 healthy weight participant (18 Kg/m2>BMI<30Kg/m2) and 20 age- and sex- matched peoples with obesity (BMI >30 Kg/m2) will be invited to a double-blinded two-way crossover MRI study, approximately 1 week apart, to assess the interplay between brain and gut to food intake.

Brain and gut MRI scans will be collected at fasted/baseline and at different time points postprandial for 120 mins using the 3T Ingenia Philips scanner. Brain measurements including resting state-fMRI, cerebral blood flow (CBF), and task-fMRI scans will be collected. During the task fMRI scan, images of high and low energy food pictures, and non-food control pictures will be presented. Food images are extensively used in fMRI studies to characterise the neural systems involved in processing the hedonic value of food as well as satiety and hunger signals. In addition to brain scans, sequences of gut scans will be collected to assess gastric volume, small bowel water content, and superior mesenteric artery (SMA) responses pre- and post-prandial. Blood samples will be collected to assess gut hormones (CCK, GLP1- PYY, ghrelin) insulin and glucose, triglycerides, free fatty acid levels at different timepoints. In addition, satiety and appetite scores will be collected using visual analogue scales. The total scan time including the fed and break times is around 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45, male and female (females will have the study days arranged during the early phase of the menstrual cycle).
* Body mass index (BMI): normal weight participants ≥ 19 and ≤ 25 Kg/m2, and obese participants > 30 Kg/m2
* Able to give voluntary written informed consent to participate in the study
* Able to understand the requirements of the study
* Apparently healthy: no medical conditions which might affect study measurements (judged by health questionnaire, and blood screening)

Exclusion Criteria:

* Any reported history of neurological or gastrointestinal disorders
* Any reported history of surgery that could affect gastrointestinal function (e.g. colectomy, small bowel resection)
* Abnormal screening procedures including depression and eat restriction
* Laboratory results that are clinically significant, including diabetes, dyslipidemia, pancreatitis, or untreated hypertension.
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury, assessed by standard MRI safety questionnaire.
* Under medication (expect aspirin/paracetamol), antibiotic or prescribed probiotic treatment in the past 12 weeks.
* Following a medically- or self-prescribed diet during the two weeks prior to the pre-study examination and until the end of the study.
* Reported weight loss or gain ≥ 10 % of bodyweight during the six months period before the pre-study examination
* Pregnancy or breastfeeding declared by candidate
* Smoking
* Left-handed assessed by handedness questionnaire. This is to control for brain's lateralisation effects (activation in one side of the brain) that may show variations between left and right handed participants.
* Participation in another clinical or research study within the previous 3 months of the study
* Cannot lie flat or exceeding the scanner bed weight limit of 250 kg.
* Poor understanding of the spoken and/or written English language

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in appetite- and satiety-related brain responses between drinks ( Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS obese) | From baseline to up to 2 hours after ingesting the drinks
  Blood oxygen level-dependent (BOLD) responses to high-calorie, low-calorie and non-food images
Changes in Cerebral blood flow between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Cerebral blood flow differences
Changes resting state brain networks between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Alterations in functional brain connectivity/networks in brain regions involved in homeostatic and hedonic brain circuits.
Changes in gastric volume between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Area Under the Curve of post-prandial gastric volumes, measured by MRI
Correlations between gut and brain responses to assess alterations in brain-gut axis between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Exploratory correlations between brain and gut responses

SECONDARY OUTCOMES:
Changes in small bowel water content between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Area Under the Curve of post-prandial small bowel water content, measured by MRI, up to 2h (AUC2h) postprandially
Changes in satiety and appetite regulators between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Area Under the Curve of post-prandial serum gut hormone (CCK, GLP-1, PYY, Ghrelin), insulin, free fatty acid, glucose, and triglyceride concentrations
Changes in satiety and appetite score (VAS) between drinks (Fat drink VS Carbohydrate drink) and across groups (Healthy weight VS Obese) | From baseline to up to 2 hours after ingesting the drinks
  Area Under the Curve for appetite (Fullness, Hunger, Prospective food consumption) post prandial 100 mm VAS scores AUC2h
Correlations between blood, brain and gut and satiety date | From baseline to up to 2 hours after ingesting the drinks
  Exploratory correlations between blood, brain and gut responses and satiety data

CONTACTS AND LOCATIONS:
Overall Officials: Sally Eldeghaidy, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
will be available upon reasonable request